CLINICAL TRIAL: NCT06671717
Title: Pralatrexate Combined With Chidamide Bridging Allogeneic Hematopoietic Stem Cell Transplantation for Refractory/Relapsed Peripheral T-cell Lymphoma
Brief Title: Pralatrexate Combined With Chidamide Bridging Allogeneic HSCT for Refractory/Relapsed Peripheral T-cell Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Ruijin Hospital (Other); Wuhan TongJi Hospital (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUPH-PTCL-001
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Relapsed Peripheral T-Cell Lymphoma; Refractory Peripheral T-Cell Lymphoma
Keywords: Allogeneic hematopoietic stem cell transplantation; Pralatrexate; Remission status before transplantation
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pralatrexate combined with Chidamide bridging allo-HSCT for Relapse/Refractory PTCL patients (Experimental): Pralatrexate combined with Chidamide bridging allo-HSCT for Relapse/Refractory PTCL patients
  Interventions: Other: Pralatrexate combined with Chidamide bridging Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Other: Pralatrexate combined with Chidamide bridging Allogeneic Hematopoietic Stem Cell Transplantation — Drug: Pralatrexate, Chidamide
  1. Pralatrexate: 30 mg/m2 intravenously (IV) administered weekly in 6-week cycles. Chidamide: 20mg, twice a week in 3-week cycles (2 weeks on treatment, 1 week off treatment)
  2. After the 6-week therapy, the patients should receive PET/CT evaluation.
  3. Patients would receive allo-HSCT if they could achieve at least PR after the first cycle of therapy. For the patients could not achieve a least PR after the first cycle of therapy, they should receive a second cycle of pralatrexate combined with chidamide. The interval between two cycles of pralatrexate combined with chidamide should be at least 1 week.
  4. After the second cycle of 6-week therapy, the patients should receive PET/CT evaluation. Patients would receive allo-HSCT if they could achieve at least SD after the second cycle of therapy. For the patients could not achieve a least SD after the second cycle of therapy, they should receive other salvage therapies.

SUMMARY:
This is a multicenter, prospective study of Pralatrexate combined with Chidamide bridging Allogeneic Hematopoietic Stem Cell Transplantation for Refractory/Relapsed Peripheral T-cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand the study, voluntarily participate in and sign on the informed consent;
* Diagnosed by histopathology Peripheral T-cell lymphoma;
* ECOG PS score 0 or 1;
* Relapsed or Refractory Peripheral T Cell Lymphoma；
* According to the 2014 version of the Lugano criteria for lymphoma, there must be at least one CT/MRI measurable lesion (measurable lymph node diameter>1.5cm; measurable extranodal lesion diameter>1.0cm)；
* Provided a written pathological/histological diagnosis report during the screening period and agreed to provide tumor tissue sections or tumor/lymph node tissue specimens for testing at the central laboratory;
* Expected survival at least 12 weeks；
* Agreed to receive treatment with Pralatrexate

Exclusion Criteria:

* NK/T-cell lymphoma;
* Achieving CR or PR after induction chemotherapies without relapse;
* Dysfunction of vital organs;
* Serious history of autoimmune diseases and immunodeficiency, including: positive for human immunodeficiency virus (HIV) antibodies; Or other acquired or congenital immunodeficiency diseases; Or have a history of organ transplantation;
* Unwilling to accept allogeneic hematopoietic stem cell transplantation;
* Undergoing other clinical studies within a month;
* Without donor for transplantation;
* Allergies to similar drugs and excipients of the research drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 1 year after transplantation | Participants will be followed for an expected average of 1 years after transplantation
  The time from the end of transplantation to progression of disease or death at 1year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Mo, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University, Institute of Hematolgoy, Beijing,, Beijing, China